CLINICAL TRIAL: NCT02061462
Title: Extracorporeal Lung Perfusion and Ventilation to Evaluate the Eligibility for Transplantation of Lungs Retrieved From Donors After Cardio-circulatory Death (DCD)
Brief Title: EVLP to Evaluate the Eligibility for Transplantation of DCD-Lungs
Acronym: EVLP-DCD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Collaborators: San Gerardo Hospital (Other)
Responsible Party: Principal Investigator, Franco Valenza, MD, Assistant Professor Anaesthesia and Intensive Care, Department of Pathophysilogy and Transplantation, Università degli Studi di Milano, Policlinico Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EVLP_2013
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Disorders Related to Lung Transplantation; Graft Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Group (No Intervention): Recipients of lungs procured from brain dead donors.
- EVLP-DCD Group (Active Comparator): Recipients of lungs procured from DCD donors, reconditioned/evaluated by EVLP
  Interventions: Procedure: EVLP-DCD Group

INTERVENTIONS:
Procedure: EVLP-DCD Group — Events: application of an open lung protective ventilatory strategy (recruitment manoeuvre, low volume-low frequency ventilation-high PEEP) to the DCD donors; procurement of lungs and cold storage on ice; reconditioning/evaluation by EVLP to assess suitability for transplantation; cold storage on ice; transplantation. Endpoints of suitability: oxygenation, respiratory mechanics, pulmonary vascular resistance, chest X-ray, fibrobronchoscopy
  Arms: EVLP-DCD Group

SUMMARY:
The procurement of organs from donors after cardiocirculatory death (DCD) is an accepted strategy to increase organ supply.

DETAILED DESCRIPTION:
Aim of the investigation: to compare the clinical outcome after transplantation of subjects receiving lungs procured from donors after cardiocirculatory death reconditioned and assessed by EVLP, with that of subjects receiving lungs procured from brain death donors.

ELIGIBILITY:
Lung donors:

* subjects with brain death according to neurological or cardiocirculatory criteria
* age below 65 yrs
* absence of massive lung contusion, aspiration, pneumonia, sepsis
* absence of infection, malignancy

Recipients:

* subjects to undergo single or bilateral lung transplantation
* informed consent to participate in the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
30 Day Mortality and Graft Survival | 30 days
  30 day mortality and graft survival is used as a standard research measure to evaluate post transplant outcome

SECONDARY OUTCOMES:
Duration of mechanical ventilation after transplantation | 30 days
ICU length of stay after transplantation | 30 days
Primary Graft Dysfunction 72 hours After Transplantation | 72 hours
  Primary Graft Dysfunction 72 hours after transplantation definition: grade 3 according to the International Society of Heart and Lung Transplantation classification

OTHER OUTCOMES:
Bronchiolitis Obliterans Syndrome (BOS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Franco Valenza, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS a' Granda - Ospedale Maggiore Policlinico, Milan, Milan, Italy